CLINICAL TRIAL: NCT02051530
Title: Mood, Serotonin and Social Interaction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Groningen (Other)
Responsible Party: Principal Investigator, Marije aan het Rot, Assistant Professor, University of Groningen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL451-09-013
Record Dates: First submitted 2014-01-24; First posted 2014-01-31 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Mood; Social Behavior
Keywords: mood; empathy; mimicry; emotional reactivity; prosody
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- tryptophan depletion first day (Experimental): tryptophan depletion on the first day. on the other day participants receive placebo.
  Interventions: Dietary Supplement: tryptophan depletion
- tryptophan depletion on day 2 (Experimental): tryptophan depletion on the second day. on the first day participants receive placebo.
  Interventions: Dietary Supplement: tryptophan depletion

INTERVENTIONS:
Dietary Supplement: tryptophan depletion — tryptophan depletion involves the ingestion of an amino acid mixture that is devoid of tryptophan. on the other day participants receive placebo, being the same mixture but including tryptophan

SUMMARY:
Rationale: Major depressive disorder (MDD) is a psychiatric disorder whose onset, severity, and duration are influenced by interpersonal factors. The serotonin system is known to influence MDD risk. Recent research has suggested that serotonin may also play a role in regulating social behaviour. Therefore, it would be interesting to study the role of serotonin in responses to social stimuli in individuals at risk for MDD.

Objective: This project aims to study how changes in serotonin alter interpersonal functioning in adults with or without a first degree family member diagnosed with MDD. The primary goal is to investigate the effect of experimentally lowered brain serotonin levels on empathic accuracy. Secondary goals are to determine how this manipulation influences verbal and non-verbal communication, cardiovascular function in a social context, and mood. An exploratory goal is to investigate how these outcomes are related to genes thought to be involved in MDD.

DETAILED DESCRIPTION:
see summary

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 yrs
* At least one first-degree family member with MDD, Family History (FH) positive, or no first and -second degree family members with MDD, FH negative
* Willingness to cooperate, to sign written informed consent

Exclusion Criteria:

* Any current or past Diagnostic and Statistical Manual (DSM) IV Axis I mood disorder, anxiety disorder, psychotic disorder, eating disorder, or somatoform disorder as determined by Structured Clinical Interview for DSM interview
* Any current substance use disorder
* Any past substance dependence
* Ongoing medical treatment for a chronic disease, particularly cancer, gastrointestinal disease, phenylketonuria, diabetes, cardiovascular disease, or disease of the liver or kidneys
* Not speaking Dutch fluently
* Current or past use of neuroleptics, sedative drugs, antidepressants etc.
* On test days, a positive urine test for drugs of abuse
* For women, initiation of hormonal contraceptive treatments 3 months prior to screening, or a positive urine test for pregnancy on test days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Empathic Accuracy | 45 minutes
  Empathic Accuracy is assessed with a computer task, approximately 6 hrs after completion of the amino acid mixture

SECONDARY OUTCOMES:
Behavioral mimicry | 10 minutes
  Behavioral mimicry is assessed in two experiments. In the first experiment, mimicry of a person in a video is assessed. In a second experiment mimicry is assessed in response to the investigators mannerisms
Emotional Prosody (EP) | 10 minutes
  EP is assessed in two experiments. In the first experiment, EP is assessed in response to a video. In a second experiment EP is assessed in a dyad with the investigator.
blood | 10 minutes
  blood is analysed for levels of tryptophan, oxytocin and cortisol
heart rate variability | 1 hour
  hrv is measured in response to emotional video clips

OTHER OUTCOMES:
Serotonin transporter polymorphism | 1 day
  From one of the blood samples collected we will isolate whole blood for DNA extraction in order to analyse the serotonin transporter polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Marije aan het Rot, Dr., Principal Investigator — University of Groningen
Locations (1):
- University Center Psychiatry, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Hogenelst K, Schoevers RA, Kema IP, Sweep FC, aan het Rot M. Empathic accuracy and oxytocin after tryptophan depletion in adults at risk for depression. Psychopharmacology (Berl). 2016 Jan;233(1):111-20. doi: 10.1007/s00213-015-4093-9. PMID 26462806